CLINICAL TRIAL: NCT02857036
Title: Characterization of Rhythmic Markers Associated With the Response to Antidepressants
Brief Title: Rhythm and Depression
Acronym: R&B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2011/120
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Depression
Keywords: rhythm; depression; antidepressant treatment
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- responder (Experimental): responder to antidepressant treatment
  Interventions: Other: rhythmic parameter recording; Behavioral: psychiatric assessment
- non responder (Experimental): non responder to antidepressant treatment
  Interventions: Other: rhythmic parameter recording; Behavioral: psychiatric assessment

INTERVENTIONS:
Other: rhythmic parameter recording — the following rhythmic parameters are recording during 48 hours: temperature, heart rate and actimetry
Behavioral: psychiatric assessment — different psychometric scales are filled in: Montgomery and Asberg depression rating scale (MADRS), Quick inventory depression scale (QIDS-C16) and Beck depression inventory (BDI)

SUMMARY:
The study aims to characterize the rhythmic parameters of unipolar depressed patients that are associated with the response to antidepressants after 6 weeks of treatment.

DETAILED DESCRIPTION:
Patients are included at the time of their hospitalization in the psychiatry unit. They perform rhythmic parameters recording within 48hours after the initiation of the antidepressant treatment. An evaluation of the evaluation of the severity of depression symptoms is performed at 2, 4 and 6 weeks after the initiation of the antidepressant treatment.

A correlation analysis will be performed with rhythmic parameters and the response to the antidepressant treatment.

ELIGIBILITY:
Inclusion Criteria:

* current unipolar major depressive disorder according to the Diagnostic ans Statistics Manual (DSM)V
* MADRS score > 25

Exclusion Criteria:

* other psychiatric disorder
* current treatment with thymoregulating agent
* clozapine treatment
* heart disease that could alter heart rate characteristics
* disease associated with fever
* shift work within 3 months before inclusion
* transmeridian travel in the preceding month
* guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
significant difference of temperature amplitude between responder and non-responder | 6 weeks
  the response to the antidepressant treatment is determined by the variation of the MADRS score between pretreatment and 6 weeks of treatment.
  the complete response is obtained when the MADRS score has at least a 50% decrease after 6 weeks.
significant difference of activity duration between responder and non-responder | 6 weeks
significant difference of RR interval of the heart rate between responder and non-responder | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Haffen, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, Doubs, France

IPD SHARING:
Plan to Share IPD: No